CLINICAL TRIAL: NCT05638373
Title: Clinical Evaluation of Shade Matching and Marginal Discoloration of One Shade Universal Resin Composite Versus Conventional Nanohybrid Resin Composite in Class IV Restorations Before and After Tooth Bleaching .
Brief Title: Shade Matching of Universal Versus Conventional Nanohybrid Resin Composites in Class IV Restorations After Bleaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nayra Mohamed Mohab El Din Hussein Mohamed, Master degree candidate, Department of Conservative Dentistry, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universal composite
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Anterior Teeth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One shade universal composite (Experimental): shade matching composite
  Interventions: Other: One shade universal composite
- Nanohybrid resin composite (Active Comparator): Conventional Nanohybrid resin composite
  Interventions: Other: Nanohybrid resin composite

INTERVENTIONS:
Other: One shade universal composite — A resin composite with new smart chromatic technology and chameleon effect. It has the ability to match the new lighter shade of the bleached teeth unlike the conventional composite
  Arms: One shade universal composite
Other: Nanohybrid resin composite — A conventional resin composite with multiple shades
  Arms: Nanohybrid resin composite

SUMMARY:
The aim of the current study is to assess the shade matching potential of single shade universal resin composite versus conventional nanohybrid resin composite in class IV restorations after bleaching

DETAILED DESCRIPTION:
The use of a dental material that can blend into the surrounding tooth structure is increasing in popularity . A new technology , smart chromatic technology , has been introduced as the shade matching composite called omnichroma . Omnichroma has the ability to match the new lighter shade of the bleached teeth unlike the conventional composite . In this study , an investigation will be done to evaluate if this new technology will help to preserve the tooth structure and be more conservative , by avoiding the removal of the old anterior restorations after bleaching

ELIGIBILITY:
Inclusion Criteria:

* Candidates must have one or more existing class IV restoration.
* Cases indicated for bleaching.
* Cooperative patient approving to participate in the trial.

Exclusion Criteria:

* Patients with severe medical conditions that might interfere with the study.
* Patients with rampant caries or xerostomia.
* Smoking.
* Patients with history of hydrogen peroxide sensitivity , periodontal inflammation.
* Lack of compliance.
* Tempromandibular joint disorders.
* Disabilities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in shade matching | Baseline, 2 days, 3, 6 and 12 months
  Modified USPHS criteria with Alpha, Bravo ,Charlie and Delta scores (Categorical)

SECONDARY OUTCOMES:
Change in Marginal discoloration | Baseline, 2 days, 3, 6 and 12 months
  Modified USPHS criteria with Alpha, Bravo, Charlie and Delta scores (Categorical)
Change in surface texture | Baseline, 2 days, 3, 6 and 12 months
  Modified USPHS criteria with Alpha, Bravo, Charlie and Delta scores (Categorical)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed El Zoheiry, prof, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ameedee AAL, Ragab H, Essam E, et al.(2016): Clinical evaluation of in-office tooth bleaching effects on three contemporary composite resins. J Dent Health Oral Disord Ther., 5(6):350-357.
- [Background] Bayne SC, Schmalz G. Reprinting the classic article on USPHS evaluation methods for measuring the clinical research performance of restorative materials. Clin Oral Investig. 2005 Dec;9(4):209-14. doi: 10.1007/s00784-005-0017-0. No abstract available. PMID 16421996
- [Background] Elzayat, G. A., Elsayed, M. E., & El Zoghby, A. (2020): Clinical Performance of Direct Anterior Composite Restorations Using Esthetic Dual-Shade versus Polychromatic Natural Layering Technique: a split mouth randomized controlled clinical trial. Brazilian Dental Science, 23(4), 12-12.
- [Background] Evans, M. B. (2020):The Visual and Spectrophotometric Effect of External Bleaching on OMNICHROMA Resin Composite and Natural Teeth. West Virginia University.
- [Background] Mohamed, M. A., Afutu, R., Tran, D., Dunn, K., Ghanem, J., Perry, R., & Kugel, G. (2020): Shade Matching Capacity of Omnichroma in Anterior Restorations. Journal of Dental Sciences., 5(1), 1-6.
- [Background] Mourouzis P, Koulaouzidou EA, Helvatjoglu-Antoniades M. Effect of in-office bleaching agents on physical properties of dental composite resins. Quintessence Int. 2013 Apr;44(4):295-302. doi: 10.3290/j.qi.a29154. PMID 23479582
- [Background] Pereira Sanchez N, Powers JM, Paravina RD. Instrumental and visual evaluation of the color adjustment potential of resin composites. J Esthet Restor Dent. 2019 Sep;31(5):465-470. doi: 10.1111/jerd.12488. Epub 2019 May 16. PMID 31095870
- [Background] Telang A, Narayana IH, Madhu KS, Kalasaiah D, Ramesh P, Nagaraja S. Effect of Staining and Bleaching on Color stability and Surface Roughness of Three Resin Composites: An in vitro study. Contemp Clin Dent. 2018 Jul-Sep;9(3):452-456. doi: 10.4103/ccd.ccd_297_18. PMID 30166843